CLINICAL TRIAL: NCT06182930
Title: The Effect of Education Given to Caregivers of Alzheimer's Patients Registered With Home Health Services on Their Knowledge and Attitudes Towards Alzheimer's Disease: Randomized Controlled Study
Brief Title: Education of Caregivers of Alzheimer's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Assoc. Prof., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ordu123456
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Education
Keywords: Alzheimer, Caregiver, Knowledge, Attitude, Education
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Within the scope of the research, caregivers will be given face-to-face training in 2 sessions, 15 days apart.
  Interventions: Other: Within the scope of the research, caregivers will be given face-to-face training in 2 sessions, 15 days apart.
- Control (No Intervention): They will receive routine home health care follow-up.

INTERVENTIONS:
Other: Within the scope of the research, caregivers will be given face-to-face training in 2 sessions, 15 days apart. — They will receive routine home health care follow-up.
  Other Names: No Intervention
  Arms: Experimental

SUMMARY:
Purpose of the Research: This study will be conducted to determine the effect of the education given to caregivers of Alzheimer's patients registered to home health services on their knowledge and attitudes towards Alzheimer's disease.

Hypotheses of the Research H01: The education given to caregivers of Alzheimer's patients registered to home health services does not affect the caregivers' level of knowledge about Alzheimer's disease.

H11: The education given to caregivers of Alzheimer's patients registered to home health services increases the caregivers' level of knowledge about Alzheimer's disease.

H02: The education given to caregivers of Alzheimer's patients registered to home health services does not affect the caregivers' attitudes towards Alzheimer's disease.

H12: The education given to caregivers of Alzheimer's patients registered to home health services positively affects the caregivers' attitudes towards Alzheimer's disease.

DETAILED DESCRIPTION:
-The number of elderly population is increasing in the world and in Turkey. Dementia increases with age. The most common type of dementia is Alzheimer's disease. As the Alzheimer's disease stage progresses, patients' dependency level in daily living activities increases and they need care support. Alzheimer's patients are usually cared for at home by family members. Caregivers may experience many difficulties in the home environment due to lack of knowledge in disease management. This study will be conducted to determine the effect of the education given to caregivers of Alzheimer's patients registered to home health services on their knowledge and attitudes towards Alzheimer's disease. The research was planned as a single-blind randomized controlled experimental study. The research will be conducted on caregivers of Alzheimer's patients registered to Giresun Province Bulancak State Hospital Home Health Services between 20 December 2023 and 20 December 2024. The population of the research will be the caregivers of Alzheimer's patients registered to Giresun Province Bulancak State Hospital Home Health Services. The sample of the research will be the caregivers of 60 patients who meet the research criteria and agree to participate in the research. The data of the study will be collected with the "Patient and Caregiver Introduction Form", "Alzheimer's Disease Information Scale" and "Dementia Attitude Scale". Necessary institutional permissions and ethics committee approval will be obtained for the research. In the research, caregivers in the experimental group will be trained about Alzheimer's disease in 2 sessions, 15 days apart, in the training hall of the hospital. No intervention will be applied to caregivers in the control group during the research. Necessary institutional permission and ethics committee approval will be obtained for the research. The analysis of the data will be done in a computer environment by an expert statistician.

ELIGIBILITY:
Inclusion Criteria:

* Those who are primarily responsible for the care of the patient diagnosed with Alzheimer's disease,
* Caring for a patient diagnosed with Alzheimer's disease for at least 6 months,
* Ages 18 and over,
* The one who is literate,
* Open to communication and collaboration,
* Caregivers who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Cannot understand and speak Turkish,
* Those with mental and cognitive retardation and
* Caregivers who do not want to continue the research will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Knowledge Scale | In the pre-test of the research, the "Alzheimer's Disease Knowledge Scale" will be administered to the caregivers by the researcher, and the "Alzheimer's Disease Knowledge Scale" will be administered again 1 month later.
  The scale developed by Carpenter et al. (2009) was adapted to Turkish by Yılmaz and Çolak (2020). The scale consists of 30 items and evaluates people's level of knowledge about Alzheimer's disease. Scale items can be answered as true or false, and participants receive one point for each item they answer correctly. The scores that can be obtained from the scale vary between 0 and 30. An increase in the score obtained from the scale indicates that the level of knowledge is high. While the difficulty index values of the scale items ranged between 0.24 and 0.75, the discrimination index was calculated above 0.10. The test-retest reliability calculated to evaluate the reliability of the scale was found to be 0.81, and the Kuder-Richardson 20 coefficient was found to be 0.74.
Dementia Attitude Scale | In the pre-test of the research, the "Dementia Attitude Scale" will be administered to the caregivers by the researcher, and the "Dementia Attitude Scale" will be administered again 1 month later.
  The scale was developed by O'Connor and McFadden in 2010 and translated into Turkish by Çetinkaya et al. Adapted from (2020). The scale was used with university students and direct care workers. During the creation of the scale, the expression "Alzheimer's disease and related diseases" was used in the scale expressions due to the terminological confusion between Alzheimer's Disease and Dementia. The scale is a 7-point Likert type, from 1 (strongly disagree) to 7 (strongly agree). 6 items of the scale, which consists of a total of 20 items, are reverse scored (2,6,8,9,16,17). As the score obtained from the scale increases, supportive and accepting attitudes increase, while exclusionary attitudes decrease. Cronbach's alpha value of the scale was found to be 0.83.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK Uğur, Asoss.Prof., Principal Investigator — Ordu Univercity
Locations (1):
- Hacer GÖK UĞUR, Ordu, Cumhuriyet Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No